CLINICAL TRIAL: NCT06483360
Title: Methane and Hydrogen Breath Test for the Diagnosis of Small Intestinal Bacterial Overgrowth
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); West China Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Chief physician, Professor, Vice president, Shanghai Jiao Tong University School of Medicine
Other Study IDs: LY2024-109-B
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Small Intestinal Bacterial Overgrowth
Keywords: Small intestinal bacterial overgrowth; Methane and hydrogen breath test; Cut-off

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The body exhales air
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate whether the positive rates of methane and hydrogen breath test were different between the experimental group and the control group.

DETAILED DESCRIPTION:
Small intestinal bacterial overgrowth (SIBO) refers to a syndrome of gastrointestinal symptoms caused by changes in the number and/or type of bacteria in the small intestine, and is considered to be secondary to changes in intestinal anatomy, slowing of intestinal motility, or abnormalities in gastrointestinal function. Clinical symptoms of SIBO are atypical, and are mainly characterized by bloating, belching, abdominal pain, diarrhea, constipation, and changes in stool shape, color, odor, and other characteristics. Since the clinical symptoms of SIBO are not specific and the clinical diagnosis criteria are not standardized, its treatment has not been given enough attention.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the experimental group:

1. Age 18-65 years old and gender;
2. Patients with functional gastrointestinal disease are characterized by abdominal symptoms (abdominal distension, early satiety, diarrhea, constipation, abdominal pain, etc.)
3. have the autonomy to complete methane and hydrogen breath testing and gastrointestinal symptom scoring independently or with medical assistance;
4. able to complete the signing of informed consent as required.

Inclusion criteria for the control group:

1. Age 18-65 years old and gender;
2. Healthy individuals without obvious typical gastrointestinal symptoms;
3. Autonomy to complete methane and hydrogen breath testing and gastrointestinal symptom scoring independently or with medical assistance;
4. Ability to complete the informed consent form as required.

Exclusion Criteria:

1. Patients whose gastroenteroscopy within one year indicated malignant tumor of digestive tract, or whose above examination proved peptic ulcer within two months;
2. A history of malignant tumors of the digestive system (not limited to the digestive tract), a history of inflammatory bowel disease, or a history of false or mechanical ileus;
3. Gastrointestinal resection, appendectomy and cholecystectomy within one year;
4. History of gastrointestinal perforation, gastrointestinal bleeding, cholangitis, acute and chronic pancreatitis within one year;
5. There is evidence of gastrointestinal tract infection (Helicobacter pylori, acute infectious enteritis);
6. History of type I diabetes and primary hypothyroidism;
7. Confirmed lactose malabsorption, lactose intolerance, and pancreatic exocrine insufficiency;
8. Within 4 weeks, a history of antibiotic administration;
9. Within 2 weeks, history of endoscopy;
10. Within 1 week, history of taking gastrointestinal stimulants, probiotics, laxatives;
11. 1 day prior to testing, eating fermentable foods (yogurt, kimchi, soy sauce, tempeh, oats, beer, etc.);
12. Not fasting 8 hours prior to testing;
13. Smoking, strenuous exercise 2 hours before and during the test;
14. Preparation for pregnancy, pregnancy, breastfeeding women, or overall poor compliance, or other conditions that the investigator believes need to be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects attending the digestive (internal) Department and physical examination department/physical examination center of each center.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Methane and hydrogen breath test results of experimental and control groups | July 1, 2024 to December 31, 2024
  To investigate whether the positive rates of methane and hydrogen breath test were different between the experimental group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-yuan Fang, MD,Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine